CLINICAL TRIAL: NCT04457752
Title: A Randomised Controlled Multicentre Clinical Trial, Evaluating the Efficacy of Dual Layer Amniotic Membrane (Artacent®) and Standard of Care Versus Standard of Care Alone in the Healing of Chronic Diabetic Foot Ulcers
Brief Title: Evaluating the Efficacy of Dual Layer Amniotic Membrane (Artacent®)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SerenaGroup, Inc. (Network)
Collaborators: Tides Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HITIDE
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Chronic Diabetic Foot Ulcers

STUDY DESIGN:
Intervention Model Description: Dual Layer Amniotic Membrane (DLAM). Artacent® Artacent® is a double layer of dehydrated amniotic membrane. The amnion is harvested from human placenta obtained during planned Caesarean sections. Tides Medical uses a proprietary process to clean and decellularize the amniotic membrane. The amnion is then folded into a bi-layer with the stromal sides facing outward. The dual layer is dried and cut into various sizes. In the final step the DLAM is terminally sterilized.
  Atracent®, like all other placental-derived products, is FDA cleared for homologous use through the 361 pathway. It is indicated for non-healing ulcers applied to a debrided, clean and uninfected ulcers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dual Layer Amniotic Membrane (DLAM) + SOC (Active Comparator): DLAM (Up to 10 weekly DLAM applications) + Standard of Care (sharp debridement, offloading, and proper moisture balance).
  Interventions: Biological: Dual Layer Amniotic Membrane (DLAM). Artacent®
- Standard of Care (No Intervention): Standard of Care: sharp debridement, offloading, and proper moisture balance.

INTERVENTIONS:
Biological: Dual Layer Amniotic Membrane (DLAM). Artacent® — Artacent® is a double layer of dehydrated amniotic membrane. The amnion is harvested from human placenta obtained during planned Caesarean sections. Tides Medical uses a proprietary process to clean and decellularize the amniotic membrane. The amnion is then folded into a bi-layer with the stromal sides facing outward. The dual layer is dried and cut into various sizes. In the final step the DLAM is terminally sterilized.
  Atracent®, like all other placental-derived products, is FDA cleared for homologous use through the 361 pathway. It is indicated for non-healing ulcers applied to a debrided, clean and uninfected ulcers.
  Arms: Dual Layer Amniotic Membrane (DLAM) + SOC

SUMMARY:
A Randomized Controlled Multicenter Clinical Trial, Evaluating the Efficacy of Dual Layer Amniotic Membrane (Artacent®) and Standard of Care versus Standard of Care alone in the healing Chronic Diabetic Foot Ulcers. Multi-center, open label, randomized controlled trial. Study is estimated to require 12 months from first subject enrolled to last subject visit.

DETAILED DESCRIPTION:
Diabetic foot ulcers (DFUs) challenge the most experienced wound care specialist. The US Wound Registry reports that only 40% of DFUs heal in 12 weeks1. Woundologists have adopted the phrase, "time is tissue." This adage reminds clinicians that the longer a DFU remains open, the greater the risk of infection, major amputation and death. The diabetic with a foot ulcer has a mortality rate of 47% which exceeds the mortality2 from most common cancers3. Beyond patient suffering, the treatment of DFUs cost the US health care system more than 15 billion dollars annually4.

In recent years, several clinical trials have demonstrated that products derived from human placental membranes promote the healing of DFUs5. Research has confirmed that growth factors present in amniotic membrane induce angiogenesis, stimulate human dermal fibroblast proliferation, and recruit stem cells important to wound repair and regeneration to the DFU6. All these factors are highly desirable properties in the healing of chronic DFUs.

A novel dual layer amniotic membrane (DLAM, Artacent™, Tides Medical. Lafayette, LA) potentially can increase the delivery of growth factors due to its double layer of amniotic membrane. A prospective case series demonstrated good healing rates in DFUs: 65% healing at 12 weeks7. The current study is the first randomized clinical trial evaluating the efficacy of DLAM in DFUs.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 18 years of age or older,
2. Subjects must have a diagnosis of type 1 or 2 Diabetes mellitus.
3. At randomization subjects must have a target ulcer with a minimum surface area of 0.7 cm2 and a maximum surface area of 20.0 cm2 measured post debridement with the Tissue Analytics photographic planimetry App.
4. The target ulcer must have been present for a minimum of 4 weeks and a maximum of 52 weeks of standard of care prior to the initial screening visit.
5. The target ulcer must be located on the foot with at least 50% of the ulcer below the malleolus.
6. The target ulcer must be full thickness without exposed bone.
7. The affected limb must have adequate perfusion confirmed by vascular assessment. Any of the following methods performed within 3 months of the first screening visit are acceptable:

   1. ABI between 0.7 and ≤ 1.3;
   2. TBI ≥ 0.6;
   3. TCOM ≥ 40 mmHg;
   4. PVR: biphasic.
8. If the subject has two or more ulcers, they must be separated by at least 2 cm. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
9. Target ulcers located on the plantar aspect of the foot must be offloaded for at least 30 days prior to randomization.
10. The subject must consent to using the prescribed off-loading method for the duration of the study.
11. The subject must agree to attend the weekly study visits required by the protocol.
12. The subject must be willing and able to participate in the informed consent process.

Exclusion Criteria:

1. A subject known to have a life expectancy of < 6 months is excluded.
2. The subject is excluded if the target ulcer is not secondary to diabetes.
3. If the target ulcer is infected or if there is cellulitis in the surrounding skin, the subject is excluded.
4. If there is evidence of osteomyelitis complicating the target ulcer, the subject is excluded.
5. A potential subject cannot have an infection in the target ulcer or in a remote location that requires systemic antibiotic therapy.
6. A subject receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of Prednisone per day or equivalent) or cytotoxic chemotherapy is excluded.
7. The topical application of steroids to the ulcer surface within one month of initial screening is not permitted.
8. A subject with a previous partial amputation on the affected foot is excluded if the resulting deformity impedes proper offloading of the target ulcer.
9. If a subject has glycated hemoglobin (HbA1c) greater than or equal to 12% within 3 months of the initial screening visit he/she is excluded.
10. The subject is excluded if the surface area measurement of the Target ulcer decreases by 40% or more during the 4-week screening phase: the 4 weeks from the initial screening visit (SV1) to the TV-1/randomization visit during which time the subject received SOC.
11. A Subject with an acute Charcot foot, or an inactive Charcot foot, that impedes proper offloading of the target ulcer is excluded.
12. Women who are pregnant or considering becoming pregnant within the next 6 months are excluded.
13. A potential subject with end stage renal disease requiring dialysis is excluded.
14. A subject who participated in a clinical trial involving treatment with an investigational product within the previous 30 days is excluded.
15. A subject who in the opinion of the investigator, has a medical or psychological condition that may interfere with study assessments is excluded.
16. A Subject treated with hyperbaric oxygen therapy or a Cellular and/or Tissue Product (CTP) in the 30 days prior to the initial screening visit is excluded.
17. A Subject is excluded if the MolecuLight Device shows a positive fluorescence image in the wound bed on TV1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Complete Wound Closure | 1-12 weeks
  - The percentage of target ulcers achieving complete wound closure in 12 weeks

SECONDARY OUTCOMES:
Percentage Wound Area Reduction | 1-12 weeks
  - Percentage wound area reduction from TV-1 to TV-13 measured weekly with digital photographic planimetry and physical examination
Adverse Events | 1-12 weeks
  The number of adverse events
Percentage of time wearing offloading boot | 1-12 Weeks
  - Compliance with a prescribed offloading boot measured as % of time wearing the boot
Pain Scale (The Pain, Enjoyment of Life and General Activity Scale). 0 = no pain , 10 = pain as bad as you can imagine | TV-1, 3 weeks, 6 weeks, 9 weeks, and 12 weeks or Final Visit
  - Change in pain in the target ulcer assessed using the PEG scale. [Time Frame: TV-1, 3 weeks, 6 weeks, 9 weeks, and 12 weeks or Final Visit]
Changes in bacterial Load | 1-12 Weeks
  - Exploratory Endpoint: changes in bacterial load measured using fluorescence imaging

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Serena, MD,FACS, Principal Investigator — Serena Group, Inc
Locations (16):
- United States (15):
  - Titan Research, Phoenix, Arizona
  - New Hope Podiatry, Los Angeles, California
  - Royal Research, Pembroke Pines, Florida
  - Pharma Research Associates, Westchester, Florida
  - Regional Infectious Disease and Infusion Center, Inc, La Grange, Georgia
  - Hoosier Foot and Ankle, Fishers, Indiana
  - Serena Group Baton Rouge, Baton Rouge, Louisiana
  - Opelousas Medical Research Consultants, LLC, Opelousas, Louisiana
  - Mount Sinai St. Luke's Hospital, New York, New York
  - Cleveland Foot and Ankle Clinic, Cleveland, Ohio
  - Heal Foundation, Tulsa, Oklahoma
  - The Foot and Ankle Wellness Center of Western Pennsylvania, Ford City, Pennsylvania
  - Armstrong County Memorial Hospital - Wound Clinic, Kittanning, Pennsylvania
  - Martin Foot and Ankle, York, Pennsylvania
  - Mt.Olympus Medical Research, Sugar Land, Texas
- Clinical Research Management Group, Coto Laurel, Puerto Rico